CLINICAL TRIAL: NCT04622046
Title: A Phase 3, Prospective, Multicenter, Open Label, 2-Part Study of the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of ALXN2060 in Japanese Participants With Symptomatic Transthyretin Amyloid Cardiomyopathy (ATTR-CM)
Brief Title: A Phase 3 Study of ALXN2060 in Japanese Participants With Symptomatic ATTR-CM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Collaborators: Eidos Therapeutics, a BridgeBio, Inc. Company (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALXN2060-TAC-302
Record Dates: First submitted 2020-11-06; First posted 2020-11-09 (Actual); Results first posted 2024-12-16 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Symptomatic Transthyretin Amyloid Cardiomyopathy
MeSH Terms: interventions — attruby

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ALXN2060 (Experimental): Participants will receive ALXN2060.
  Interventions: Drug: ALXN2060

INTERVENTIONS:
Drug: ALXN2060 — ALXN2060 tablets will be administered twice daily at a dose of 800 milligrams.
  Other Names: AG10; Acoramidis

SUMMARY:
This prospective study is designed to evaluate the efficacy, safety, and tolerability of ALXN2060 (also known as AG10), as well as to establish its pharmacokinetic and pharmacodynamic profile in Japanese participants with symptomatic ATTR-CM administered on a background of stable heart failure therapy.

DETAILED DESCRIPTION:
Participants will receive ALXN2060 for 12 months (Part A). Following the last visit (Month 12) of Part A, participants will continue the study in Part B, which will last for an additional 18 months (30 months from Day 1), during which all participants will continue to receive oral treatment with ALXN2060. Following completion of Month 30 assessments in Part B, participants will be offered the opportunity to continue to receive ALXN2060 in the Extension Period, which will last until ALXN2060 is approved in Japan or for up to 24 additional months, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Established diagnosis of ATTR-CM with either wild-type TTR or a variant TTR genotype.
2. History of heart failure evidenced by at least 1 prior hospitalization for heart failure or clinical evidence of heart failure without prior heart failure hospitalization manifested by signs or symptoms of volume overload or elevated pressures or heart failure symptoms that required or requires ongoing treatment with a diuretic.
3. New York Heart Association Class I-III symptoms due to ATTR-CM.
4. On stable doses of cardiovascular medical therapy.
5. Completed ≥ 150 meters on the 6MWT on 2 tests prior to Day 1.
6. Left ventricular (LV) wall (interventricular septum or LV posterior wall) thickness ≥ 12 millimeters.
7. Biomarkers of myocardial wall stress: N-terminal pro-brain-type natriuretic pep (NT-proBNP) level ≥ 300 picograms/milliliter (pg/mL).

Exclusion Criteria:

1. Acute myocardial infarction, acute coronary syndrome or coronary revascularization, or experienced stroke or transient ischemic attack within 90 days prior to screening.
2. Hemodynamic instability at screening.
3. Likely to undergo heart transplantation within a year of screening.
4. Current treatment with marketed drug products and other investigational agents for the treatment of ATTR-CM.
5. Current treatment with calcium channel blockers with conduction system effects (for example, verapamil, diltiazem). The use of dihydropyridine calcium channel blockers is allowed.
6. Confirmed diagnosis of light-chain (AL) amyloidosis.
7. Biomarkers of myocardial wall stress: NT-ProBNP ≥ 8,500 pg/mL.
8. Measure of kidney function, estimated glomerular filtration rate by Modification of Diet in Renal Disease formula < 30 mL/minute/1.73 meters squared.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-11-13 (Actual); Primary Completion 2023-11-08 (Actual); Study Completion 2025-08-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- Japan (11):
  - Research Site, Bunkyō City
  - Research Site, Fukuoka
  - Research Site, Kumamoto
  - Research Site, Kurume-shi
  - Research Site, Matsumoto-shi
  - Research Site, Nagoya
  - Research Site, Nankoku-shi
  - Research Site, Sagamihara-shi
  - Research Site, Sapporo
  - Research Site, Shinjuku-ku
  - Research Site, Suita-shi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ALXN2060-TAC-302&attachmentIdentifier=4fcbc7a5-80cf-43d9-8c9e-88f9e62c3866&fileName=ALXN2060-TAC-302_CSR_Synopsis_21_Mar_2024_signed_redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Data presented in this results posting are for analyses up to the Month 30 visit (Intervention Period). The Extension Period of the study is ongoing. Data for the Extension Period will be reported once the study has completed.
Groups:
- ALXN2060: Participants received ALXN2060 twice daily (bid) for 12 months (Part A). Following the Month 12 visit, participants continued to receive ALXN2060 bid for an additional 18 months (up to 30 months from Day 1, [Part B]). Following the completion of Month 30 assessments, participants were offered the opportunity to continue into the Extension Period for up to 30 additional months or until ALXN2060 could be provided via an Alexion post study access program (as allowed by local laws and regulations), whichever occurred first. The Extension Period of the study is ongoing.
Period: Intervention Period
Arm/Group | ALXN2060
Started | 25
Received at Least 1 Dose of Study Drug | 25
Completed | 22
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 2
Period: Extension Period
Arm/Group | ALXN2060
Started | 21 (One participant did not proceed to the Extension Period after completing the Intervention Period.)
Completed | 0
Not Completed | 21
Not completed — Ongoing in the Extension Period | 21

BASELINE CHARACTERISTICS:
Population: Full Analysis Set, which included all participants who have received at least 1 dose of ALXN2060.
Arm/Group | ALXN2060
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.5 (6.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 25
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Part A: Change From Baseline To Month 12 Of Treatment In Distance Walked During The Six-minute Walk Test (6MWT)
Description: The 6MWT measures how far a participant can walk in 6 minutes. Change from baseline was calculated as the difference between the distance walked during the 6MWT at 12 months and the distance walked during the 6MWT at baseline. To determine the baseline, at least 2 6MWTs were conducted > 24 hours to ≤ 3 weeks apart prior to the first dose of ALXN2060. The baseline 6MWT is the average of the total distance walked by participants for the 2 qualifying 6MWTs that met all the protocol-defined criteria. Least squares mean change from baseline data were adjusted for baseline measures and visits.
Time Frame: Baseline, Month 12
Population: Measured in the Full Analysis Set, which included all participants who have received at least 1 dose of ALXN2060. Number of participants analyzed = number of participants evaluable for the outcome measure at the specified timepoint.
Measure: Least Squares Mean (Standard Error); unit: meters
Arm/Group | ALXN2060
Number analyzed (Participants) | 23
meters | -3.86 (9.182)

2. Primary Outcome: Parts A and B: Number of Cardiovascular (CV)-Related Hospitalizations Over A 30-month Period
Description: CV-related hospitalization was defined as the mean number of CV-related hospitalizations per participant per year over a 30-month period. CV-related hospitalizations were also reported as adverse events and were reviewed and adjudicated by an independent Clinical Events Committee (CEC).
Time Frame: 30 months
Population: Measured in the Full Analysis Set, which included all participants who have received at least 1 dose of ALXN2060.
Measure: Mean (95% Confidence Interval); unit: CV-related hospitalizations
Arm/Group | ALXN2060
Number analyzed (Participants) | 25
CV-related hospitalizations | 0.1329 [0.0511 to 0.3457]

3. Secondary Outcome: Parts A and B: Change From Baseline In Distance Walked During The 6MWT
Description: The 6MWT measures how far a participant can walk in 6 minutes. Change from baseline was calculated as the difference between the distance walked during the 6MWT at specified timepoints and the distance walked during the 6MWT at baseline. To determine the baseline, at least 2 6MWTs were conducted > 24 hours to ≤ 3 weeks apart prior to the first dose of ALXN2060. The baseline 6MWT is the average of the total distance walked by participants for the 2 qualifying 6MWTs that met all the protocol-defined criteria. Least squares mean change from baseline data were adjusted for baseline measures and visits.
Time Frame: Baseline, Months 6, 9, 18, 24 and 30
Population: Measured in the Full Analysis Set, which included all participants who have received at least 1 dose of ALXN2060. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure. "Number analyzed" = participants evaluable for this outcome measure at the specified timepoint.
Measure: Least Squares Mean (Standard Error); unit: meters
Arm/Group | ALXN2060
Number analyzed (Participants) | 25
meters
  Month 6 | -29.54 (9.316)
  Month 9: number analyzed (Participants) | 23
  Month 9 | -23.12 (11.610)
  Month 18: number analyzed (Participants) | 19
  Month 18 | -26.27 (12.532)
  Month 24: number analyzed (Participants) | 22
  Month 24 | -24.89 (8.534)
  Month 30: number analyzed (Participants) | 22
  Month 30 | -36.20 (10.798)

4. Secondary Outcome: Parts A and B: Change From Baseline In The Kansas City Cardiomyopathy Questionnaire Overall Score (KCCQ-OS)
Description: The KCCQ is a 23-item questionnaire developed to measure health status and health-related quality of life in participants with heart failure. Items include heart failure symptoms, impact on physical and social functions, and how their heart failure impacts their quality of life. The overall summary score ranged from 0-100, with higher scores indicating better health status. Data presented are for change from baseline to specified timepoints. Least squares mean change from baseline data were adjusted for baseline measures and visits.
Time Frame: Baseline, Months 6, 9, 12, 18, 24 and 30
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | ALXN2060
Number analyzed (Participants) | 25
scores on a scale
  Month 6 | 0.94 (2.779)
  Month 9: number analyzed (Participants) | 23
  Month 9 | -1.73 (3.291)
  Month 12: number analyzed (Participants) | 23
  Month 12 | 2.71 (2.766)
  Month 18: number analyzed (Participants) | 21
  Month 18 | -5.34 (3.747)
  Month 24: number analyzed (Participants) | 22
  Month 24 | -0.68 (3.029)
  Month 30: number analyzed (Participants) | 22
  Month 30 | -6.97 (3.755)

5. Secondary Outcome: Parts A and B: Number of Participants With Treatment-emergent Adverse Events (AEs), Serious Adverse Events (SAEs) and AEs Leading to Treatment Discontinuation
Description: A treatment-emergent AE was defined as any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention that occurred after first dose. A treatment-emergent SAE was defined as any untoward medical occurrence that resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent disability/incapacity, or was a congenital anomaly/birth defect that occurred after first dose. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Up to Month 30
Population: Measured in the Safety Set, which included all participants who have received at least 1 dose of ALXN2060.
Measure: Count of Participants; unit: Participants
Arm/Group | ALXN2060
Number analyzed (Participants) | 25
Participants
  Treatment-emergent AE | 25
  Treatment-emergent SAE | 12
  AEs Leading to Treatment Discontinuation | 2

6. Secondary Outcome: Parts A and B: Change From Baseline In Serum Transthyretin (TTR) Concentration
Description: Least squares mean change from baseline derived from with visits and baseline serum TTR as a covariate. Other covariates were included as needed.
Time Frame: Baseline, pre-dose on Days 14, 28 and Months 3, 6, 9, 12, 15, 18, 21, 24, 27 and 30
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: milligrams (mg)/deciliter (dL)
Arm/Group | ALXN2060
Number analyzed (Participants) | 24
milligrams (mg)/deciliter (dL)
  Day 14, Predose | 9.73 (0.886)
  Day 28, Predose | 9.13 (1.256)
  Month 3, Predose | 10.64 (1.056)
  Month 6, Predose: number analyzed (Participants) | 23
  Month 6, Predose | 9.61 (0.847)
  Month 9, Predose: number analyzed (Participants) | 23
  Month 9, Predose | 11.16 (0.744)
  Month 12, Predose: number analyzed (Participants) | 22
  Month 12, Predose | 11.80 (1.157)
  Month 15, Predose: number analyzed (Participants) | 22
  Month 15, Predose | 10.79 (1.347)
  Month 18, Predose: number analyzed (Participants) | 22
  Month 18, Predose | 10.12 (1.253)
  Month 21, Predose: number analyzed (Participants) | 22
  Month 21, Predose | 9.23 (0.704)
  Month 24, Predose: number analyzed (Participants) | 22
  Month 24, Predose | 11.06 (0.848)
  Month 27, Predose: number analyzed (Participants) | 22
  Month 27, Predose | 9.57 (1.020)
  Month 30, Predose: number analyzed (Participants) | 21
  Month 30, Predose | 9.36 (1.280)

7. Secondary Outcome: Parts A and B: Change From Baseline In TTR Stabilization
Description: TTR stabilization was measured using fluorescent probe exclusion (FPE). Data presented are for change from baseline in FPE percentage stabilization.
Time Frame: Baseline, Pre-dose Days 14, 28 and Months 3, 6, 9, 12, 15, 18, 21, 24, 27 and 30
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: percentage stabilization
Arm/Group | ALXN2060
Number analyzed (Participants) | 24
percentage stabilization
  Day 14, Predose | 97.15 [94.45 to 100.05]
  Day 28, Predose | 97.29 [95.16 to 99.66]
  Month 3, Predose | 99.09 [95.24 to 102.64]
  Month 6, Predose: number analyzed (Participants) | 23
  Month 6, Predose | 98.56 [94.20 to 104.44]
  Month 9, Predose: number analyzed (Participants) | 23
  Month 9, Predose | 96.47 [94.07 to 101.73]
  Month 12, Predose: number analyzed (Participants) | 22
  Month 12, Predose | 100.89 [99.95 to 102.51]
  Month 15, Predose: number analyzed (Participants) | 22
  Month 15, Predose | 97.65 [96.30 to 100.03]
  Month 18, Predose: number analyzed (Participants) | 22
  Month 18, Predose | 96.75 [94.40 to 101.00]
  Month 21, Predose: number analyzed (Participants) | 22
  Month 21, Predose | 101.30 [99.80 to 103.00]
  Month 24, Predose: number analyzed (Participants) | 22
  Month 24, Predose | 102.60 [98.20 to 104.80]
  Month 27, Predose: number analyzed (Participants) | 22
  Month 27, Predose | 102.65 [101.00 to 105.60]
  Month 30, Predose: number analyzed (Participants) | 21
  Month 30, Predose | 95.60 [91.60 to 103.60]

8. Primary Outcome: All-cause Mortality (ACM) Over A 30-month Period
Description: ACM was assessed as time from the date of first initiation of study treatment to the date of death during a 30-month period, and was analyzed using Kaplan-Meier analysis. Data are reported for the number of participants with ACM over the 30-month period.
Time Frame: 30 months
Population: Measured in the Full Analysis Set, which included all participants who have received at least 1 dose of ALXN2060.
Measure: Count of Participants; unit: Participants
Arm/Group | ALXN2060
Number analyzed (Participants) | 25
Participants | 0

ADVERSE EVENTS:
Time Frame: Up to Month 30
Description: All-cause mortality is reported for all enrolled participants. Serious and other adverse events are reported for the Safety Set, which included all participants who have received at least 1 dose of ALXN2060.
Arm/Group | ALXN2060
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 12/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ALXN2060 (N=25)
Atrial fibrillation (Cardiac disorders) | 1
Atrioventricular block complete (Cardiac disorders) | 1
Cardiac discomfort (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Cardiac failure chronic (Cardiac disorders) | 1
Sinus arrest (Cardiac disorders) | 1
Sinus node dysfunction (Cardiac disorders) | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Large intestine polyp (Gastrointestinal disorders) | 2
Appendicitis perforated (Infections and infestations) | 1
Bacterial prostatitis (Infections and infestations) | 1
Pneumonia pneumococcal (Infections and infestations) | 1
Blood creatine phosphokinase MB increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Soft tissue mass (Musculoskeletal and connective tissue disorders) | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Device dislocation (Product Issues) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ALXN2060 (N=25)
Anaemia (Blood and lymphatic system disorders) | 2
Atrial flutter (Cardiac disorders) | 2
Cardiac failure (Cardiac disorders) | 2
Palpitations (Cardiac disorders) | 2
Vertigo (Ear and labyrinth disorders) | 2
Dry eye (Eye disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 3
Malaise (General disorders) | 2
Pyrexia (General disorders) | 5
COVID-19 (Infections and infestations) | 4
Cystitis (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 6
Limb injury (Injury, poisoning and procedural complications) | 2
Blood creatinine increased (Investigations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 2
Gout (Metabolism and nutrition disorders) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Carpal tunnel syndrome (Nervous system disorders) | 2
Haematuria (Renal and urinary disorders) | 4
Renal impairment (Renal and urinary disorders) | 4
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-09-11): https://cdn.clinicaltrials.gov/large-docs/46/NCT04622046/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-27): https://cdn.clinicaltrials.gov/large-docs/46/NCT04622046/SAP_001.pdf